CLINICAL TRIAL: NCT02489721
Title: PICC and Midline Related Complications: A Multicenter Observational Study
Brief Title: Major Complications Related to PICC and Midline Insertion
Acronym: PICC/MIDLINE
Status: Completed | Type: Observational
Sponsor: Azienda Ospedaliera S. Maria della Misericordia (Other)
Responsible Party: Principal Investigator, Livia Pompei, Medical Doctor, Azienda Ospedaliera S. Maria della Misericordia
Other Study IDs: PICC/MIDLINE1
Record Dates: First submitted 2015-06-30; First posted 2015-07-03 (Estimated); Last update posted 2020-01-13 (Actual); Status verified 2020-01

CONDITIONS: Upper Extremity Deep Vein Thrombosis
Keywords: peripherally inserted central venous catheter; depp vein thrombosis; related blood stream infections; midline
MeSH Terms: conditions — Upper Extremity Deep Vein Thrombosis | interventions — Catheterization, Peripheral

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: PICC and Midline — Peripherally inserted central venous catheter

SUMMARY:
Most important peripherally inserted central catheter (PICC) and Midline complications are thrombosis and catheter related blood stream infections. No large prospective observational study are present in literature about these topics. The aim of this multicenter prospective observational study is to analyze all the complications due to PICC and Midline insertion.

DETAILED DESCRIPTION:
A PICC line is a Peripherally Inserted Central Catheter. It is long, small, flexible tube that is inserted into a peripheral vein, typically in the upper arm, and terminates in a large vein in the chest to obtain a central intravenous access. A Midline catheter is similar to a PICC, but it is shorter in length (about 25 cm) and is inserted into a large vein in the upper arm, terminating not beyond the axillary vein. Midline catheters offer a longer dwell time and better hemodilution than the short peripheral IV catheters.The use of PICC and Midline has been increasing in outpatient and inpatient settings. Factors driving this increased use include their ease of insertion due to the placement into a peripheral vein-a safer approach-with the benefit of a central tip location appropriate for any osmolarity and pH infusions, a low reported incidence of infection, a better patient comfort, a durable venous access, and an easier nursing management in outpatient setting. PICC placement under ultrasound guidance can be carried out with no iatrogenic, mechanical complications associated with central venous catheter insertion in the neck or chest (pneumothorax, hemothorax etc…). Despite their many advantages, recent data suggest that PICCs are associated with venous thromboembolism. The incidence of symptomatic thrombosis ranges from 1.9% to 8.4% and it increases to 75% considering also the asymptomatic one. The risk factors that predispose a patient to the development of a thrombotic complication are: the caliber of the device (≥5Fr), the position of the catheter tip, the insertion of the PICC in a paretic limb, a history of venous thrombosis, the residence time of the device and the presence of an oncological pathology. The second major complication due to the PICC insertion is the catheter related blood stream infection (CRBSI). The incidence of PICC-BSI in literature ranges from 2.0 per 1000 catheter days to 3.1 per 1000 catheter days. This disparity stems from the fact that there is no single definition of catheter infection. Multiple factors associated with patient and catheter care have been identified has having an increased risk of CRBSI and are amenable to preventive measures. Independent risk factors for PICC BSIs included congestive heart failure, intrabdominal perforation, Clostridium difficile infection, recent chemotherapy, presence of tracheostomy, and type of catheter (double or tri lumen). Limited data exists regard prospective observational study on deep vein thrombosis and CRBSI related to PICC and Midline insertion, including the different calibers of the device and the presence of single or multiple lumen.

The investigators designed a multicenter prospective observational study to determine the incidence of deep vein thrombosis, related/associated catheter blood stream infections and the incidence of all the minor complications due to PICC and Midline insertion.

ELIGIBILITY:
Inclusion Criteria:

• all patients aged 18-90 years (oncological, malignancy hematology, medical, surgical and critically ICU patients) in whom it was determined that PICC/Midline insertion was indicated.

Exclusion Criteria:

* renal insufficiency whose creatinine level was greater than 3.0 mg/dL or who were undergoing hemodialysis,
* preexisting bacteremia (ie, existing positive blood cultures that had not been repeated with negative results);
* preexisting venous thrombosis or known hypercoagulable states (such as protein C or S deficiency, Antithrombin deficiency, lupus anticoagulant);
* axillary lymphonodi dissection or alteration of lymphatic drainage;
* PICC and/or Midline insertion in a paretic arm;
* patients who had been previously enrolled in the trial.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will be conducted in all the patients undergoing PICC or Midline catheter insertion which fall in the inclusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 547 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2020-01 (Actual); Study Completion 2020-01 (Actual)

PRIMARY OUTCOMES:
Prevalence of deep venous thrombosis (DVT) occurring after the PICC placement in all patients | 2 years

SECONDARY OUTCOMES:
Prevalence of infections related catheter | 2 years
Prevalence of other complications such as phlebitis, occlusion, malposition | 2 years
Reason of the catheter removal | 2 years
Prevalence of the same complications Midline related | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Livia Pompei, MD, Principal Investigator — AOU Santa Maria della Misericordia; Giorgio Della Rocca, MD, Study Director — AOU Santa Maria della Misericordia
Locations (1):
- AOU Santa Maria della Misericordia, Udine, Italy

REFERENCES:
- [Result] Greene MT, Flanders SA, Woller SC, Bernstein SJ, Chopra V. The Association Between PICC Use and Venous Thromboembolism in Upper and Lower Extremities. Am J Med. 2015 Sep;128(9):986-93.e1. doi: 10.1016/j.amjmed.2015.03.028. Epub 2015 May 1. PMID 25940453
- [Result] Chopra V, Fallouh N, McGuirk H, Salata B, Healy C, Kabaeva Z, Smith S, Meddings J, Flanders SA. Patterns, risk factors and treatment associated with PICC-DVT in hospitalized adults: A nested case-control study. Thromb Res. 2015 May;135(5):829-34. doi: 10.1016/j.thromres.2015.02.012. Epub 2015 Feb 21. PMID 25726426